CLINICAL TRIAL: NCT01076010
Title: An Extension Treatment Protocol for Subjects Who Have Participated in a Phase 3 Study of Tivozanib vs. Sorafenib in Renal Cell Carcinoma (Protocol AV-951-09-301).
Brief Title: An Extension Treatment Protocol for Subjects Who Have Participated in a Study of Tivozanib Versus Sorafenib in Kidney Carcinoma (Protocol AV-951-09-301).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-09-902; 2009-015987-32 (EudraCT Number)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — tivozanib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sorafenib crossover to tivozanib. (Experimental): The subjects who failed sorafenib (had Response Evaluation Criteria in Solid Tumors [RECIST] - defined progressive disease) on the parent protocol AV-951-09-301 will be offered tivozanib hydrochloride on Protocol AV- 951-09-902.
  Interventions: Drug: Tivozanib; Drug: Sorafenib
- First line tivozanib. (Experimental): The subjects who were randomized to tivozanib (continued from the parent Protocol AV-951-09-301) and demonstrated clinical benefit and acceptable tolerability in Protocol AV-951-09-301.
  Interventions: Drug: Tivozanib
- First line sorafenib. (Active Comparator): The subjects who were randomized to sorafenib (continued from the parent Protocol AV-951-09-301) and demonstrated clinical benefit and acceptable tolerability were to be offered long-term access to sorafenib.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Tivozanib — Tivozanib capsules, administered orally, on a dosing schedule of 3 weeks of treatment (beginning on Day 1) followed by 1 week off treatment. One cycle was defined as 4 weeks of treatment.
  Arms: First line tivozanib.; Sorafenib crossover to tivozanib.
Drug: Sorafenib — Sorafenib tablets, 400 mg twice daily, administered orally for 4 weeks (1 cycle = 4 weeks). One cycle was defined as 4 weeks of treatment. Cycles were repeated every 4 weeks.
  Arms: First line sorafenib.; Sorafenib crossover to tivozanib.

SUMMARY:
Open-label, multi-center extension treatment protocol to allow access to tivozanib and sorafenib for subjects who have participated on the AV-951-09-301 protocol. Eligible subjects who were randomized to receive sorafenib on AV-951-09-301 and had documented progression of disease will receive a tivozanib dose of 1.5 mg/day. Eligible subjects who were randomized to tivozanib or sorafenib in AV-951-09-301, and displayed clinical benefit and acceptable tolerability to treatment, will continue to receive tivozanib or sorafenib at the same dose and schedule as in AV-951-09-301.

DETAILED DESCRIPTION:
This is an extension treatment protocol to allow access to tivozanib or sorafenib for subjects enrolled on AV-951-09-301(parent protocol). Subjects who failed sorafenib on the parent protocol will be offered tivozanib. Subjects who were randomized to tivozanib, and demonstrated clinical benefit and acceptable tolerability will be offered long-term access to tivozanib. Subjects who were randomized to sorafenib, and demonstrated clinical benefit and acceptable tolerability will be offered long-term access to sorafenib. Subjects who continue receiving sorafenib on this protocol and progress will be allowed to cross-over to tivozanib.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have participated on Protocol AV-951-09-301, and must meet either of the following bulleted criteria:

   * Demonstrated disease progression per RECIST during treatment with sorafenib, OR
   * Demonstrated clinical benefit [complete response (CR), partial response (PR), or stable disease (SD) per RECIST] and acceptable tolerability after treatment with tivozanib or sorafenib on protocol AV-951-09-301.
2. Eastern Cooperative Oncology Group performance status ≤ 2 and life expectancy ≥ 3 months.
3. If female and of childbearing potential, documentation of negative pregnancy test prior to enrollment.
4. Ability to give written informed consent

Exclusion Criteria:

1. Newly identified central nervous system (CNS) malignancies or documented progression of CNS metastases; subjects will be allowed only if the CNS metastases have been adequately treated with radiotherapy or surgery. For subjects receiving steroid therapy for allowed steroid maintenance therapy.
2. Duration since last dose on Protocol AV-951-09-301:

   1. For subjects continuing tivozanib or sorafenib (subjects who demonstrated clinical benefit and acceptable tolerability during treatment with tivozanib or sorafenib on protocol AV-951-09-301): more than 2 weeks since last dose of tivozanib or sorafenib.
   2. For subjects initiating tivozanib (ie demonstrated disease progression during treatment with sorafenib): more than 4 weeks since last dose of sorafenib. Subjects demonstrating disease progression due to CNS metastasis will be allowed up to 8 weeks since last dose of sorafenib in order to complete treatment for CNS metastasis.
3. Inadequate recovery from any prior surgical procedure or major surgical procedure within 4 weeks prior to administration of first dose of study drug.
4. Any of the following hematologic abnormalities:

   * Hemoglobin < 9.0 g/dL
   * Absolute neutrophil count < 1500 per mm3
   * Platelet count < 75,000 per mm3
   * Prothrombin time or Partial thromboplastin time >1.5 × upper limit of normal (ULN)
5. Any of the following serum chemistry abnormalities:

   * Total bilirubin > 1.5 × ULN (or > 2.5 × ULN for subjects with Gilbert's syndrome)
   * Aspartate aminotransferase or alanine aminotransferase > 2.5 × ULN (or > 5 × ULN for subjects with liver metastasis)
   * Alkaline phosphatase > 2.5 × ULN (or > 5 × ULN for subjects with liver or bone metastasis)
   * Creatinine > 2.0 × ULN
   * Proteinuria > 3+ by urinalysis or urine dipstick
6. If female, pregnant or lactating.
7. Sexually active pre-menopausal female subjects (and female partners of male subjects) must use adequate contraceptive measures, while on study and for at least 50 days after the last dose of study drug. Sexually active male subjects must use adequate contraceptive measures, while on study and for at least 90 days after the last dose of study drug. All fertile male and female subjects,and their partners,must agree to use a highly effective method of contraception. Effective birth control includes (a) Intrauterine device plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). (Note: Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are not considered effective for this study).
8. Uncontrolled hypertension: systolic blood pressure > 150 mmHg or diastolic blood pressure >100 mmHg on 2 or more antihypertensive medications, documented on 2 consecutive measurements taken at least 24 hours apart.
9. Unhealed wounds (including active peptic ulcers).
10. Serious/active infection or infection requiring parenteral antibiotics.
11. Life-threatening illness or organ system dysfunction compromising safety evaluation.
12. Psychiatric disorder, altered mental status precluding informed consent or necessary testing.
13. Inability to comply with protocol requirements.
14. Treatment with another anti-cancer therapy or participation in another interventional protocol (excluding AV-951-09-301).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (75):
- United States (5):
  - Site 185, Los Angeles, California
  - Site 184, Orlando, Florida
  - Site 182, Minneapolis, Minnesota
  - Site 186, New York, New York
  - Site 187, Dallas, Texas
- Bulgaria (5):
  - Site 403, Plovdiv
  - Site 404, Sofia
  - Site 400, Sofia
  - Site 401, Varna
  - Site 402, Veliko Tarnovo
- Site 110, Montreal, Quebec, Canada
- Chile (2):
  - Site 122, Santiago
  - Site 123, Temuco
- Site 411, Prague, Czechia
- Site 133, Saint-Herblain, France
- Hungary (3):
  - Site 423, Budapest
  - Site 421, Kaposvár
  - Site 422, Pécs
- India (8):
  - Site 156, Ahmedabad, Gujarat
  - Site 151, Nashik, Maharashtra
  - Site 153, Pune, Maharashtra
  - Site 191, Jaipur, Rajasthan
  - Site 152, Vellore, Tamil Nadu
  - Site 158, Lucknow, Uttar Pradesh
  - Site 150, Kolkata, West Bengal
  - Site 154, Delhi
- Italy (3):
  - Site 160, Arezzo
  - Site 161, Pavia
  - Site 162, Roma
- Poland (7):
  - Site 432, Bialystok
  - Site 434, Bydgoszcz
  - Site 431, Gdansk
  - Site 435, Olsztyn
  - Site 433, Poznan
  - Site 430, Warsaw
  - Site 436, Warsaw
- Romania (5):
  - Site 444, Brasov
  - Site 441, Bucharest
  - Site 440, Bucharest
  - Site 443, Bucharest
  - Site 442, Timișoara
- Russia (18):
  - Site 459, Ufa, Bashkortostan Republic
  - Site 451, Chelyabinsk
  - Site 452, Kazan'
  - Site 454, Moscow
  - Site 453, Moscow
  - Site 458, Moscow
  - Site 460, Moscow
  - Site 461, Moscow
  - Site 462, Moscow
  - Site 450, Nizhny Novgorod
  - Site 456, Obninsk
  - Site 467, Omsk
  - Site 463, Pyatigorsk
  - Site 457, Rostov-on-Don
  - Site 466, Saint Petersburg
  - Site 465, Saint Petersburg
  - Site 464, Yaroslavl
  - Site 455, Yekaterinburg
- Serbia (5):
  - Site 480, Belgrade
  - Site 481, Belgrade
  - Site 482, Belgrade
  - Site 484, Kamenitz
  - Site 483, Niš
- Ukraine (9):
  - Site 491, Chernihiv
  - Site 498, Dniproperovsk
  - Site 492, Dniproperovsk
  - Site 493, Donetsk
  - Site 496, Donetsk
  - Site 490, Ivano-Frankivsk
  - Site 494, Kharkiv
  - Site 497, Uzhhorod
  - Site 495, Zaporizhia
- United Kingdom (2):
  - Site 170, Cambridge
  - Site 172, Leicester

REFERENCES:
- See also: Related Info — http://www.aveopharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 55 sites in 14 countries. Study Period from 24 May 2010 (First Subject Dosed) to 04 July 2014 (Last Subject Last Visit).
Pre-assignment Details: All participants underwent inclusion and exclusion criteria assessment and all eligible subjects signed the informed consent before undergoing any study related procedures. All the study assessments were performed as per the schedule of assessment.
Period: Overall Study
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Started | 161 | 88 | 28
Completed | 36 | 49 | 26
Not Completed | 125 | 39 | 2
Not completed — Death | 15 | 1 | 0
Not completed — Adverse Event | 7 | 2 | 0
Not completed — Progressive disease | 90 | 30 | 1
Not completed — Lack of Efficacy | 4 | 0 | 0
Not completed — Treatment Interruption for > 2 Weeks | 0 | 1 | 0
Not completed — Significant Surgical Procedure | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Noncompliance | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1
Not completed — Other | 5 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib | First Line Sorafenib | Total
Number analyzed (Participants) | 161 | 88 | 28 | 277
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 58 | 17 | 195
  >=65 years | 41 | 30 | 11 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 33 | 9 | 88
  Male | 115 | 55 | 19 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 0 | 9
  Not Hispanic or Latino | 154 | 84 | 28 | 266
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 156 | 87 | 28 | 271
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Subjects Received Treatment in Each Treatment Arm
Description: Number of days subjects received treatment who were from Protocol AV-951-09-301 who either continued on tivozanib in this trial (subjects with first-line experience on tivozanib treatment), who crossed over from sorafenib to tivozanib in this trial (crossover subjects) participated in, and who continued on sorafenib in this trial (subjects with first-line experience on sorafenib treatment). Subjects could be discontinued due to unacceptable toxicities or clinical or documented PD
Time Frame: From enrollment to until all subjects discontinue (due to documented progressive disease [PD] or unacceptable toxicities) or until 3 years after the first subject was enrolled in Protocol AV-951-09-902
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
Days
  Duration of Treatment | 290 (234.37) | 325.3 (137.79) | 369.4 (107.6)
  Total Days Receiving Drug | 222.36 (181.722) | 241.0 (105.928) | 368.14 (107.946)

2. Primary Outcome: Number of Cycles Subjects Received Treatment in Each Treatment Arm
Description: Number of cycles subjects received who were from Protocol AV-951-09-301 who either continued on tivozanib in this trial (subjects with first-line experience on tivozanib treatment), who crossed over from sorafenib to tivozanib in this trial (crossover subjects) participated in, and who continued on sorafenib in this trial (subjects with first-line experience on sorafenib treatment). Subjects could be discontinued due to unacceptable toxicities or clinical or documented PD
Time Frame: From enrollment to until all subjects discontinue (due to documented PD or unacceptable toxicities) or until 3 years after the first subject was enrolled in Protocol AV-951-09-902
Measure: Mean (Standard Deviation); unit: Number of cycles started
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
Number of cycles started | 10.6 (8.36) | 11.8 (4.85) | 13.2 (3.83)

3. Primary Outcome: Total Dose Administered to Subjects in Each Treatment Arm (mg)
Description: The total dose administered to subjects who were from Protocol AV-951-09-301 who either continued on tivozanib in this trial (subjects with first-line experience on tivozanib treatment), who crossed over from sorafenib to tivozanib in this trial (crossover subjects) participated in, and who continued on sorafenib in this trial (subjects with first-line experience on sorafenib treatment). Subjects could be discontinued due to unacceptable toxicities or clinical or documented PD
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
mg | 318.84 (256.241) | 344.58 (152.131) | 244014.29 (116816.715)

4. Primary Outcome: Average Daily Dose Administered to Subjects in Each Treatment Arm
Description: The average daily dose administered to subjects who were from Protocol AV-951-09-301 who either continued on tivozanib in this trial (subjects with first-line experience on tivozanib treatment), who crossed over from sorafenib to tivozanib in this trial (crossover subjects) participated in, and who continued on sorafenib in this trial (subjects with first-line experience on sorafenib treatment). Subjects could be discontinued due to unacceptable toxicities or clinical or documented PD
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
mg/day | 1.46 (0.121) | 1.40 (0.196) | 651.47 (225.410)

5. Primary Outcome: Relative Dose Intensity (RDI) of Treatment Administered to Subjects in Each Treatment Arm
Description: RDI is defined as 100% times the actual dose intensity divided by the intended dose intensity. The RDI of subjects who were from Protocol AV-951-09-301 who either continued on tivozanib in this trial (subjects with first-line experience on tivozanib treatment), who crossed over from sorafenib to tivozanib in this trial (crossover subjects) participated in, and who continued on sorafenib in this trial (subjects with first-line experience on sorafenib treatment). Subjects could be discontinued due to unacceptable toxicities or clinical or documented PD
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
percentage of dose | 95.21 (9.393) | 91.12 (14.762) | 80.60 (28.603)

6. Primary Outcome: Number of Subjects With Adverse Events
Description: Number of subjects with Treatment-Related Adverse Events (AEs) as assessed by Common Terminology Criteria for Adverse Events v3.0
Time Frame: From enrollment assessed up to 3 years of treatment or until follow-up (up to 30 days end-of-trial visit after treatment discontinuation), whichever occurs earlier
Population: Number of subjects with adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
Participants
  AE | 124 | 85 | 28
  Any AE of Grade 3 or Higher | 77 | 55 | 19
  Any Treatment-Related AE | 86 | 76 | 27
  Any Treatment-Related Any Treatment AE ≥ Grade 3 | 39 | 35 | 15
  Any AE With Outcome of Death | 21 | 3 | 0
  Any treatment-Related AE With Outcome of death | 1 | 1 | 0
  Any serious adverse event (SAE) | 49 | 17 | 4
  Any treatment-related SAE | 7 | 7 | 2
  AE leading to study drug discontinuation (AEDC) | 19 | 4 | 0
  Any treatment-related AEDC | 3 | 0 | 0
  AE leading to study drug interruption | 27 | 26 | 12
  Treatment-related AE - study drug interruption | 13 | 17 | 10
  AE Leading to Study Drug Dose Reduction | 11 | 11 | 10
  Treatment related AE - Study Drug Dose Reduction | 9 | 11 | 10

7. Secondary Outcome: Number of Subjects With Objective Response Rate (ORR) Who Continued Treatment With Tivozanib or Sorafenib and Who Received Tivozanib After Failure of Sorafenib
Description: ORR is defined as the proportion of subjects with confirmed complete response (CR) or confirmed partial response (PR) according to RECIST (Version 1.0), relative to the total population of dosed subjects. CR is disappearance of all target and non-target lesions and normalization of tumor marker levels. At least a 30% decrease in the sum of the loading dose (LD) of target lesions, taking as reference the baseline sum LD. To allow long-term access to sorafenib for subjects who participated in Protocol AV-951-09-301 (NCT01030783), and demonstrated clinical benefit and acceptable tolerability to sorafenib.
Time Frame: From Day 1 to the end of treatment (EOT) Visit, approximately every 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
Participants
  Overall Confirmed Objective Response Rate | 29 | 49 | 16
  Overall Unconfirmed Objective Response Rate | 43 | 55 | 16

8. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from the first documentation of objective tumor response (confirmed CR or confirmed PR) according to RECIST (Version 1.0) to the first documentation of objective tumor progression or to death due to any reason. DR was calculated for the subgroup of subjects with a confirmed objective tumor response (PR or CR). CR is Disappearance of all target and non-target lesions and normalization of tumor marker levels. PR is At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Number of subjects with disease progression or death and censored endpoints were summarized and statistical analysis were performed for duration of response.
Time Frame: From the first documentation of objective tumor response to the first documentation of objective tumor progression, assessed up to treatment discontinuation or to death due to any reason or maximum up to 3 years, whichever occurs earlier
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 29 | 49 | 16
Participants
  Subjects who had disease progression or died | 10 | 11 | 0
  Subjects with censored endpoints | 19 | 38 | 16
Statistical Analysis 1: Comparison: Sorafenib Crossover to Tivozanib; Test type: Other; 25% Quartile (months) = 8.0, 95% CI 2-sided [4.4 to 12.9]
Statistical Analysis 2: Comparison: Sorafenib Crossover to Tivozanib; Test type: Other; 50% Quartile (months) = 15.2, 95% CI 2-sided [lower limit 11.1] (DR was only summarized for subjects who had an objective tumor response. Upper limit of confidence interval could not be determined.)
Statistical Analysis 3: Comparison: First Line Tivozanib; Test type: Other; 25% Quartile (months) = 12.9, 95% CI 2-sided [lower limit 5.6] (DR was only summarized for subjects who had an objective tumor response. Upper limit of confidence interval could not be determined.)

9. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the date of first dose of study drug to the first documentation of objective tumor progression or death due to any reason, whichever occurred first. For the crossover subjects and subjects with first-line experience on tivozanib treatment, the timeframe for PFS assessment started from the date of first dose of tivozanib in the AV-951-09-902 study. For subjects with first-line experience on sorafenib treatment, the timeframe for PFS assessment started from the date of first dose of sorafenib in the AV-951-09-902. Number of subjects with disease progression or death was summarized and statistical analysis were performed for PFS.
Time Frame: From the date of first dose of study drug (tivozanib or sorafenib) in the AV-951-09-902 study to the first documentation of objective tumor progression or death due to any reason or maximum up to 3 years, whichever occurred first
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
Participants
  Subjects who had disease progression or died | 108 | 35 | 1
  Subjects with censored endpoints | 53 | 53 | 27
Statistical Analysis 1: Comparison: Sorafenib Crossover to Tivozanib; Test type: Other; 25% Quartile (months) = 3.6, 95% CI 2-sided [1.9 to 5.2]
Statistical Analysis 2: Comparison: Sorafenib Crossover to Tivozanib; Test type: Other; 50% Quartile (months) = 11.0, 95% CI 2-sided [7.3 to 12.7]
Statistical Analysis 3: Comparison: Sorafenib Crossover to Tivozanib; Test type: Other; 75% Quartile (months) = 20.9, 95% CI 2-sided [lower limit 16.5] (For the subjects in each treatment arm, PFS is calculated from the first dose date of the respective study drugs. Upper limit of confidence interval could not be determined.)
Statistical Analysis 4: Comparison: First Line Tivozanib; Test type: Other; 25% Quartile (months) = 7.2, 95% CI 2-sided [3.5 to 9.2]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study drug (tivozanib or sorafenib) date on this study to date of death due to any cause. Number of subjects died or alive was summarized and statistical analysis were performed for OS.
Time Frame: From the date of first dose of study drug (tivozanib or sorafenib) in the AV-951-09-902 study to death due to any reason or maximum up to 3 years, whichever occurred first
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib. | First Line Sorafenib.
Number analyzed (Participants) | 161 | 88 | 28
Participants
  Died | 78 | 10 | 0
  Alive | 83 | 78 | 28
Statistical Analysis 1: Comparison: Sorafenib Crossover to Tivozanib; Test type: Other; 25% Quartile (months) = 8.2, 95% CI 2-sided [6.0 to 12.1]
Statistical Analysis 2: Comparison: Sorafenib Crossover to Tivozanib; Test type: Other; 50% Quartile (months) = 21.6, 95% CI 2-sided [17.0 to 27.6]
Statistical Analysis 3: Comparison: Sorafenib Crossover to Tivozanib; Test type: Other; 75% Quartile (months) = 30.7, 95% CI 2-sided [lower limit 28.8] (For the subjects in each treatment arm, OS is calculated from the first dose date of the respective study drugs. Upper limit of confidence interval could not be determined.)

ADVERSE EVENTS:
Time Frame: From enrollment assessed up to 3 years of treatment or until follow-up (up to 30 days end-of-trial visit after treatment discontinuation), whichever occurs earlier
Description: An AE was defined as any unintended or undesirable, noxious, or pathological change, compared to pre-existing conditions, experienced by a patient during the clinical study or the follow-up period, regardless of relationship to study drug
Groups:
- Sorafenib Crossover to Tivozanib: The subjects who failed sorafenib (had RECIST-defined progressive disease) on the parent protocol will be offered tivozanib hydrochloride.
Arm/Group | Sorafenib Crossover to Tivozanib | First Line Tivozanib | First Line Sorafenib
Serious Adverse Events (participants affected / at risk) | 49/161 | 17/88 | 4/28
Other Adverse Events (participants affected / at risk) | 87/161 | 82/88 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib Crossover to Tivozanib (N=161) | First Line Tivozanib (N=88) | First Line Sorafenib (N=28)
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 0
Death (General disorders) | 2 | 1 | 0
Multi-organ failure (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0
Myxoedema (Endocrine disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Delusional disorder, somatic type (Psychiatric disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
cataract (Eye disorders) | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Salivary gland mass (Gastrointestinal disorders) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib Crossover to Tivozanib (N=161) | First Line Tivozanib (N=88) | First Line Sorafenib (N=28)
Hypertension (Vascular disorders) | 41 | 44 | 16
Diarrhoea (Gastrointestinal disorders) | 22 | 35 | 12
Fatigue (General disorders) | 21 | 20 | 3
Asthenia (General disorders) | 20 | 20 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 21 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 13 | 2
Decreased appetite (Metabolism and nutrition disorders) | 9 | 11 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 16 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 3
Nausea (Gastrointestinal disorders) | 0 | 21 | 0
Weight increased (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 21 | 9
Headache (Nervous system disorders) | 0 | 14 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 11 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 11 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 10 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 10 | 4
Proteinuria (Renal and urinary disorders) | 0 | 10 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 9 | 3
Hypothyroidism (Endocrine disorders) | 0 | 9 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 9 | 0
Vomiting (Gastrointestinal disorders) | 0 | 9 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 8 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 7 | 0
Amylase increased (Investigations) | 0 | 6 | 0
Lipase increased (Investigations) | 0 | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 5 | 0
Insomnia (Psychiatric disorders) | 0 | 5 | 0
Oedema peripheral (General disorders) | 0 | 5 | 0
alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Blood phosphorus decreased (Investigations) | 0 | 0 | 5
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 2
Lipase increased (Investigations) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 2
Rash pustular (Infections and infestations) | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No